CLINICAL TRIAL: NCT04939857
Title: Effect of Trimetazidine on Radiotherapy-induced Heart Damage in Lung Tumor Patients Treated With Stereotactic Body Radiotherapy.
Brief Title: Effect of Trimetazidine on Radiotherapy-induced Heart Damage.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKU Third Hospital
Record Dates: First submitted 2021-05-27; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Cardiotoxicity
Keywords: Trimetazidine, Radiation-induced heart damage, GLS
MeSH Terms: conditions — Cardiotoxicity | interventions — Trimetazidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Trimetazidine was given 2 weeks before radiotherapy, 20 mg each time, three times a day for 3 months.
  Interventions: Drug: Trimetazidine
- control group (No Intervention): No intervention

INTERVENTIONS:
Drug: Trimetazidine — The experimental group will be treated with trimetazidine, and the control group will not be intervened
  Arms: experimental group

SUMMARY:
This is a randomized controlled trial. 80 patients with thoracic radiotherapy will be included. Participants will be randomly divided into experimental group or control group. Before radiotherapy, echocardiography, 2D STE, CK, CK-MB, cTnT, NT-proBNP, electrocardiogram (ECG), and hs-CRP will be detected. During subsequent follow-up, echocardiography, 2D STE, CK, CK-MB, cTnT, NT-proBNP, ECG, and hs-CRP will be collected at every follow-up time.

DETAILED DESCRIPTION:
This is a randomized controlled trial. 80 patients with thoracic radiotherapy will be included in Peking University Third Hospital from May 15, 2021 to August 31, 2022. Participants will be randomly divided into experimental group or control group. Before radiotherapy, echocardiography, 2D STE, CK, CK-MB, cTnT, NT-proBNP, electrocardiogram (ECG), and hs-CRP will be detected. All participants will be followed up after completion of RT, 3 months after RT, 6 months after RT, and 12 months after RT. During subsequent follow-up, echocardiography, 2D STE, CK, CK-MB, cTnT, NT-proBNP, ECG, and hs-CRP will be collected at every follow-up time.

ELIGIBILITY:
Inclusion Criteria:

* lung tumor patients; 18-80 years old; will be treated by stereotactic body radiotherapy

Exclusion Criteria:

* Prior radiotherapy; ACS; heart failure (NYHA III-IV); arrhythmia requiring intervention; echocardiographic images that could not be satisfactorily obtained; significant valvular heart disease (defined as more than mild valvular regurgitation or stenosis).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-25 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
global longitudinal strain-A parameter of two dimensional speckle tracking echocardiography | pre-radiotherapy, 12 months after radiotherapy
  The primary outcome of the trial was a decrease in global longitudinal strain ≥10%.

SECONDARY OUTCOMES:
Rate of major adverse cardiovascular events | pre-radiotherapy, after completion of radiotherapy, 3 months after radiotherapy, 6 months after radiotherapy, and 12 months after radiotherapy
  Proportion of patients with major adverse cardiovascular events (MACE) in total participants. MACE was defined as unstable angina, new arrhythmia, acute myocardial infarction, heart failure, valvular heart disease, acute pericarditis, and cardiac death in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zhu, doctor, Study Chair — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No